CLINICAL TRIAL: NCT07153562
Title: Effect of Liuzijue Qigong Exercises on Ventilatory Function in Post Stroke Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aia Muhammad Ibrahem, assistant lecturer of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 012/005865
Record Dates: First submitted 2025-08-17; First posted 2025-09-04 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Ventilatory Function; Functional Capacity; Motor Function; Sleep Quality; Quality of Life
Keywords: liuzijue qigong; ventilatory function; stroke; elderly
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Stroke

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be assigned randomly into two groups of equal number . the randomization will be performed by computerized randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liuzijue Qigong (Experimental): 35 patients will perform : Liuzijue exercise for 20 minutes, 5 times per week, Beside conventional rehabilitation exercises, 3 sessions per week, 45-60 minutes per session, for 12 successive weeks.
  Interventions: Other: liuzijue qigong exercises; Other: conventional rehabilitation treatment
- Conventional rehabilitation (Active Comparator): 35 patients will do only conventional rehabilitation exercises, 3 sessions per week, 45-60 minutes per session, for 12 successive weeks.
  Interventions: Other: conventional rehabilitation treatment

INTERVENTIONS:
Other: liuzijue qigong exercises — Liuzijue qigong exercise for 20 minutes, 5 times per week, for 12 successive weeks.
  Arms: Liuzijue Qigong
Other: conventional rehabilitation treatment — conventional rehabilitation exercises, 3 sessions per week, 45-60 minutes per session, for 12 successive weeks.

SUMMARY:
to investigate the effect of Liuzijue Qigong exercises on ventilatory function in post stroke elderly patients.

DETAILED DESCRIPTION:
70 post stroke patients their ages ranges from 60 to 70 years old, randomly assigned into two groups: Study group (A) that consists of 35 patients (18 women &17 men) who perform Liuzijue exercise, 5 sessions per week, 20 minutes per session. and conventional rehabilitation treatment 3 sessions per week, 45-60 minutes per session, for 12 successive weeks.

Control group (B) that consists of 35 patients (18 women &17 men) in which patients receive just the conventional exercise program, 3 sessions per week, 45-60 minutes per session, for 12 successive weeks.

During the study, the participants receive study information form, instructions and signed the consent form.

ELIGIBILITY:
Inclusion criteria:

All patients included in this study met the following criteria:

1. Subject people of both sexes (18 women, and 17 men).
2. All patients had unilateral stroke.
3. Their age ranged from 60 to 80 years old.
4. Stroke onset was from 6 to 1 months.
5. Medically stable subjects.
6. Non-smoker subjects.
7. Ability to understand and follow simple verbal instructions.

Exclusion criteria:

Patients who experienced or had one or more of the following were excluded from the study:

1. Patients with severe acute illness.
2. Chronic unstable pulmonary and/or cardiac disease.
3. Impaired level of consciousness and evidence of gross cognitive problems.
4. Patients undergo chemotherapy.
5. Active hemoptysis, untreated pneumothorax, recent esophageal surgery.
6. Recent oral, facial or skull trauma / surgery, acute sinusitis, epistaxis, hemodynamic instability.
7. Current Smokers.
8. Patients had a severe psychological disorder.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
PFT | 3 MONTHS
  Spirometer to measure Forced expiratory volume in 1 second (FEV1), in liters
PFT | 3 months
  Spirometer to measure Forced vital capacity (FVC), in liters
PFT | 3 months
  Spirometer to measure maximum voluntary ventilation (MVV), in liters per minute
PFT | 3 months
  Spirometer to measure Predicted Forced expiratory volume in 1 second
PFT | 3 months
  Spirometer to measure predicted forced vital capacity
PFT | 3 MONTHS
  Spirometer to measure FEV1/ FVC

SECONDARY OUTCOMES:
aerobic capacity and endurance | 3 MONTHS
  The six minute walk test Is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity
motor function | 3 MONTHS
  The simplified FMA ( Fugl-Meyer Assessment ) for the assessment of motor function. The scale has a total score of 100, which is divided into motor function evaluation of the upper and lower limbs, among which the upper limb score is 56 and the lower limb score is 44. Each item has a 3-point rating, and a higher score indicates better motor function. The classification of its dysfunction is as follows: < 50 = severe dyskinesia; 50-84 = significant dyspraxia; 85-95 = moderate dyskinesia; 96-99 = mild dyskinesia; and 100 = normal
quality of daily life | 3 MONTHS
  The MBI ( Modified Barthel Index )to evaluate the quality of daily life. The scale is divided into ten items and evaluated on the basis of patients' functional status. The 10 items are eating, bathing, grooming, dressing, controlling bowel movements, controlling urination, toileting, bed and chair transfer, walking on flat ground, and going up and down stairs. The total score is 100 points. The classification of dysfunction is as follows: 100 points = self-care; 61-99 = mild dysfunction; 41-60 = moderate dysfunction; and ≤ 40 = severe dysfunction. The lower the MBI score, the more independent the patients are and the worse their daily living ability
sleep quality | 3 MONTHS
  The PSQI (Pittsburgh sleep quality index) consists of 19 separate items that collectively create 7 components, resulting in a total global score. A lower score indicates better sleep quality

CONTACTS AND LOCATIONS:
Overall Officials: Azza Abdelaziz Abdelhady, Professor of Physical Therapy, Study Director — faculty of physical therapy
Locations (1):
- Faculty of Physical Therapy, Dokki, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No